CLINICAL TRIAL: NCT05637177
Title: Support of Healthy Ageing: Using Educational and Psychosocial In-terventions to Maintain Mental Health, for Prevention and Timely Diagnosis of Depression, Anxiety, and Cognitive Disorders of Older Adults in a Community
Brief Title: Preventive Intervention to Promote Healthy Ageing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ostrava (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: NU21-09-00067
Record Dates: First submitted 2022-11-24; First posted 2022-12-05 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Preventive Intervention
Keywords: Mental health; quality of life; anxiety; depression; population ageing
MeSH Terms: conditions — Psychological Well-Being; Anxiety Disorders; Depression | interventions — Music Therapy; Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cognitive behavioral therapy (CBT) (Experimental): We used the "Aging Wisely" program for seniors living in the community, which uses elements of CBT and is specifically designed for older people over the age of 65 living in the community who may be in a worried, anxious or depressed mood. The program focuses on psychoeducation to manage these feelings. Seniors learn to change the ways they think and behave that maintain depression and anxiety. The sessions include education on the process of aging, coping with loneliness, improving sleep, coping with worry and avoidance, coping with loss and death. During the sessions, participants learn to track mood, motivation to change, goal setting, planning pleasant activities, identifying thoughts, working with useless thoughts, and practice techniques to replace useless thoughts. The last two sessions are dedicated to assertiveness and communication, and preventing recurrence of problems.
  Interventions: Behavioral: Anging Wisely
- Reminiscence therapy (Experimental): Reminiscence is a method of working with memories. Remembering has an irreplaceable place in every person's life. It is a natural activity that can encourage people, make them aware of their own achievements, different moments in life, point out their value, promote self-esteem and contribute to the development of relationships. Self-remembering is a natural form of cognitive stimulation.
  Interventions: Behavioral: Reminiscence therapy
- Music therapy (Experimental): The aim of music therapy is to optimize the quality of life, and to improve psychological, social, communication, emotional and mental health and well-being. Music therapy brings psychological and physical relaxation, reduces stress, improves mood, alleviates anxiety, improves memory and attention, develops and facilitates communication, enables self-expression. For this purpose, a number of activities are used, such as listening to music, singing, playing simple rhythmic instruments, playing the body and a number of other activities that will be carried out with seniors as part of the intervention.
  Interventions: Behavioral: Music therapy
- memory training (Experimental): Cognitive training is targeted and structured exercise of cognitive functions (learning, memory, attention, speech, visual-spatial functions, ability to solve problems, plan or manage various tasks and correctly recognize one's surroundings). Regular exercise of cognitive abilities can create a cognitive reserve that can delay the potential aggravation of problems in memory or attention and improve quality of life.
  The content of the intervention will be activities developing cognitive functions (primarily memory, attention, imagination, spatial orientation and decision-making speed), practical training and motivation for long-term regular strengthening of cognitive functions using the comprehensive training program MENTEM.
  Interventions: Behavioral: Cognitive training
- creation of educational modules (mental health, neural diseases …) (Experimental): Educational activities will focus on disease prevention in three main directions - cardiovascular diseases, mental health and neurological diseases. Educational activities will take place within the University of the Third Age LF OU.
  Interventions: Behavioral: Educational activities

INTERVENTIONS:
Behavioral: Anging Wisely — The program includes 11 meetings of two hours in a group of up to eight people. The sessions are held weekly. Each lesson is given a homework assignment. A total of 10 groups will take place.
  Arms: Cognitive behavioral therapy (CBT)
Behavioral: Music therapy — Music therapy sessions are held once a week for 60 minutes for 12 weeks. The maximum number of participants per group is 12. A total of 10 groups will be implemented.
  Arms: Music therapy
Behavioral: Reminiscence therapy — Reminiscence therapy sessions are held once a week for 60 minutes for 12 weeks. The maximum number of participants per group is 10. A total of 5 groups will be implemented.
  Arms: Reminiscence therapy
Behavioral: Cognitive training — Intervention "cognitive training" will take place once a week for 45 minutes for 20 weeks. Seniors can choose from two options: 1. group training full-time or home training (online) using the comprehensive training program MENTEM.
  Arms: memory training
Behavioral: Educational activities — Interventions in educational activities will run for one academic year. In total, seniors will attend 16 lectures in each educational module. The lectures will run 1 x 14 days for 90 minutes.
  Arms: creation of educational modules (mental health, neural diseases …)

SUMMARY:
The aim of the project is the support of healthy ageing of older adults in acommunity. Efficient educational and psychosocial intervention will besuggested and verified to prevent anxiety, depression, and cognitivedisorders of selected older adults, to im-prove their self-esteem,meaningfulness of life, sense of coherence, quality of life, and attitudes toold age. Correlations among anxiety, depression, cognitive functions, andcertain psychosocial aspects will be analyzed.

DETAILED DESCRIPTION:
The main objective of the project is to determine the efficiency ofeducational pro-grams and psychosocial interventions to maintain mentalhealth, to prevent and timely diagnose any depression, anxieties, andcognitive disorders in older adults living in a community. Furthermore, theaim is to ascertain the incidence of depression, anxiety, and cognitivedisorders in these older adults and its correlation to the assessment of lifemeaningfulness, self-respect, attitudes to old age and ageing, and the levelof social support. An intervention study will be carried out. A preventionprogram will be for-mulated based on the individual needs of older adults asidentified in the focus groups. Selected interventions will be performed in apresent form (face to face) as well as distance form (e-Health) and will runat least for 6 months. The assessment of anxiety, depression, cognitivefunctions, and other psychosocial aspects will be done before theinterventions start, when they finish, and 3 months after that. Based on-quantitative analysis, there will be evaluated the efficiency of the providedinterven-tion with respect to depression, anxiety, cognitive function, andpsychosocial aspects (attitudes to old age, self-esteem, the sense ofcoherence, quality of life, level of social support). Older adults in thecentrum for prevention and support healthy ageing in the community will beincluded in the research sample. Based on the findings, recommen-dations will be formulated regarding the selected interventions used in communi-tycare.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 60 years
* living at home in Moravian-Silesian region
* consent with partici-pation in the study
* no dementia diagnosis.

Exclusion Criteria:

* dementia diagnosis

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of depression: The Geriatric Depression Scale - GDS | 12 weeks
  The Geriatric Depression Scale may be used with healthy, medically ill, and mild to moderately cognitively impaired older adults. It has been extensively used incommunity, acute care, and long-term care settings. A Short Form GDS consisting of 15 questions was developed in 1986. The total score of the Geriatric Depression Scale can ranged from 0 to 15 points, and higher score indicates more depression symptoms. Scores of 0-4 are considered normal, 5-8 indicate mild depression; 9-11 indicate moderate depression; and12-15 indicate severe depression.
Assessment of anxiety: Geriatric Anxiety Inventory - GAI | 12 weeks
  The Geriatric Anxiety Inventory Scale consists of 20 "Agree/Disagree" items designed to assess the typical common anxiety symptoms. The total score of the Geriatric Anxiety Inventory Scale can ranged from 0 to 20 points, and higher score indicates more anxiety.
Assessment of cognitive functioning: Montreal Cognitive Assessment - MoCA | 12 weeks
  The MoCA evaluates different types of cognitive abilities. Theseinclude - orientation, short-term memory, executivefunction/visuospatial ability (language abilities, abstraction, animalnaming, attention), clock-drawing test. Scores on the Montreal Cognitive Assessment range from 0 to 30, with a score of 26 and higher generally considered normal. The scoring breakdown is as follows: visuospatial and executivefunctioning (5 points), animal naming (3 points), attention (6 points), language (3 points), abstraction (2 points), delayed recall (5 points), orientation (6 points), Test MoCA makes it possible to identify sooner the early cognitive disorders, because it evaluates one's memory in detail and analyzes the executive functions.
Assessment of quality of life: OPQOL-CZ-20 (Older People's Quality of Life Questionnai-re). | 12 weeks
  The Older People's Quality of Life Questionnaire (OPQoL-brief) consisted of 13 statements, with the participants being asked to indicate the extent to which they agree with each statement by selecting one of five possible options ("strongly disagree", "disagree", "neither agree nor disagree", "agree" and "strongly agree"). The range in the original version is based on the principle of point allocation (1-5). The items are summed to provide a total OPQoL-brief score. The total score of Older People's Quality of Life Questionnaire ranges from 13 to 65 and higher scores indicate better quality of life. The OPQoL-brief questionnaire also includes a preliminary single item on global quality of life. This single item is not scored with the OPQOL, it is coded as very good to very bad.
Assessment of the sense of coherence: The Sense of Coherence Scale - SOC-13 | 12 weeks
  The short form of the Sense of Coherence Scale -SOC-13 scale consists of 13 items that comprise three components: comprehensibility (to which 5 items contribute), manageability (4 items), and meaningfulness (4 items). The respondents indicate agreement or disagreement on a 7-category semantic differential scale with two anchoring responses tailored to the content of each item. The total score of the Sense of Coherence Scale can range from 13 to 91, and a higher score indicates higher sense of coherence.
Assessment of Life satisfaction: Life Satisfaction Index for the Third Age - Short Form - LSITA-SF | 12 weeks
  The Life Satisfaction Index for the Thirds Age - Short form questionnaire contains 12 items with options on the 6-point Likert scale: Strongly Disagree (6), Disagree (5), Somewhat Disagree (4), Somewhat Agree (4), Agree (2), and Strongly Agree (1). The total scores of the The Life Satisfaction Index for the Thirds Age - Short form questionnaire range from 12 to 72. Higher scores mean lower life satisfaction.
Assessment of self-esteem: Rosenberg Self-Esteem Scale - RSES | 12 weeks
  Rosenberg Self-Esteem Scale - RSES is a 10-item Likert type scale, with items answered on a four-point scale: from Strongly Agree (SA) toStrongly Disagree (SD). The total scores of the Rosenberg Self-Esteem Scale rank from 0 to 25 points. Score from 15 to 25 shows normal self-esteem and score of less than 15 shows low self-esteem. TheRosenberg Self-Esteem Scale, a widely used self-report instrument forevaluating individual self-esteem, was investigated using itemresponse theory.
Assessment of attitudes to ageing: Attitudes to Ageing Questionnaire - AAQ | 12 weeks
  The 24 items of the Attitudes to Ageing Questionnaire scale are scored on a five-point Likert scale (1 = strongly disagree, 5 = strongly agree). It consists of three broaddimensions of ageing: 1. physical functioning (8 items including health,dynamics, vitality, exercising), 2. psychological growth (8 items, whichreflect explicit gains in relation to self and others; the positive focus ofageing, life orientation, connection with "wisdom" and "fruits of life",coping, acceptance, communication with young generation), 3.psychosocial losses (8 items, when old age is primarily described as anegative experience including losses, deficiency, exclusion, loss ofindependence, depression, and loneliness). Each factor has eight questions with domains returning minimum scores of 8 and maximum of 40. Higher score indicates better attitudes to ageing.
Assessment of social support: Social Support Questionnaire - Short Form (SSQ6) | 12 weeks
  This instrument has 6 items that measure perceived social support. Foreach of the 6 items, respondents indicate the number of peopleavailable to provide support in each of 6 areas and then rate theoverall level of satisfaction with the support given in each of the areas. The total scores of the Social support Questionnaire rank from 0 to 6 points. Higher score indicates more social support.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ostrava, Ostrava, Česká Republika, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] Pachana NA, Byrne GJ, Siddle H, Koloski N, Harley E, Arnold E. Development and validation of the Geriatric Anxiety Inventory. Int Psychogeriatr. 2007 Feb;19(1):103-14. doi: 10.1017/S1041610206003504. PMID 16805925
- [Background] Laidlaw K, Power MJ, Schmidt S; WHOQOL-OLD Group. The Attitudes to Ageing Questionnaire (AAQ): development and psychometric properties. Int J Geriatr Psychiatry. 2007 Apr;22(4):367-79. doi: 10.1002/gps.1683. PMID 17051535
- [Background] Bowling A, Hankins M, Windle G, Bilotta C, Grant R. A short measure of quality of life in older age: the performance of the brief Older People's Quality of Life questionnaire (OPQOL-brief). Arch Gerontol Geriatr. 2013 Jan-Feb;56(1):181-7. doi: 10.1016/j.archger.2012.08.012. Epub 2012 Sep 19. PMID 22999305
- [Derived] Buzgova R, Bobcikova K, Kozakova R, Zelenikova R. The Czech version of the life satisfaction index for the third age-short form (LSITA-SF12): Psychometric properties. Int J Older People Nurs. 2023 Jul;18(4):e12541. doi: 10.1111/opn.12541. Epub 2023 Apr 24. PMID 37092730
- See also: Heissler R, Kopeček M, Pachana NA, Franková V, Štěpánková Georgi H. Geriatric Anxiety Inventory (GAI) and its short form GAI-SF: Czech normative study. Cesk Psychol. 2018;62(5):462-476. ISSN 0009-062X — http://cspsych.psu.cas.cz/result.php?id=1032
- See also: Antonovsky, A. Unravelling the mystery of health. How people manage stress and stay well. New York: Jossey Bass Publisher; 1987. 1st ed. 218 pp. ISBN 9781555420284 — https://searchworks.stanford.edu/view/1260798
- See also: Rosenberg M. Society and the adolescent self-image. Princeton, NJ: Princeton University Press, 1965. 326 p — https://www.academia.edu/19813736/Rosenberg_M_Society_and_the_adolescent_self_image_Princeton_NJ_Princeton_University_Press_1965_326_p